CLINICAL TRIAL: NCT05287698
Title: The Effect of Cold Vapor on Sore Throat and Dysphagia in the Early Postoperative Period After Suspension Laryngoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Dr. Özlem İbrahimoğlu, Assisstant Professor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IstanbulMU11
Record Dates: First submitted 2022-03-02; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Sore Throat; Dysphagia; Surgery
Keywords: Sore throat; Dysphagia; Laryngoscopy; Nursing Care
MeSH Terms: conditions — Pharyngitis; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Patients who were hospitalized for suspension laryngoscopy and met the sample selection criteria will be included in the experimental and control groups by block randomization method using the random numbers table on the computer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold vapor group (Experimental): Cold vapor will be applied to the experimental group patients for 15 minutes in the recovery room. For the study, Nebtime UN600A Ultrasonic Nebulizer Device will be used to apply cold steam to the patients which used in the hospital and calibrated (https://elmaslarmedikal.com.tr/urunler/nebtime-un600a-ultrasonik-nebulizator/). The parameters to be set on the device for the cold vapor to be applied to the patients in the early postoperative period will be vapor intensity level 5 (1-10), air blowing intensity 5 (1-10), heater intensity 1 (+10C), and timer 15 minutes. The patients will be evaluated by the researchers in terms of sore throat and dysphagia before and 15 minutes after the cold vapor application in the recovery room and at the 6th, 12th, and 24th hours after the cold vapor application in the postoperative service.
  Interventions: Other: Cold vapor
- Control group (No Intervention): Patients in the control group will receive standard care that includes all medical and non-medical treatments in the hospital. Nursing care, which is routinely applied to patients in the postoperative period, both in the recovery room and in the service, will be continued within the standard care. The patients will be evaluated by the researchers in terms of sore throat and dysphagia when they come to the recovery room and at the 6th,12th, and 24th hours after the surgery in the postoperative service.

INTERVENTIONS:
Other: Cold vapor — Before surgery, socio-demographic data of the patients, ASA and Mallampati scores, sore throat level, and dysphagia level will be recorded. After surgery, patients will be evaluated in the recovery room for their suitability to participate in the study with the Ramsay sedation scale and the Modified Aldrete Scale. Cold vapor will be applied to the patients for 15 minutes in the recovery room during the postoperative period. The parameters to be set on the device for the cold vapor to be applied to the patients in the early postoperative period will be vapor intensity level 5, air blowing intensity 5, heater intensity 1 (+10C), and timer 15 minutes. The patients will be evaluated by the researchers in terms of sore throat and dysphagia before and 15 minutes after the cold vapor application in the recovery room and at the 6th, 12th, and 24th hours after the cold vapor application in the postoperative service.
  Arms: Cold vapor group

SUMMARY:
Suspension laryngoscopy (SL) is a surgical procedure that is widely applied in the diagnosis and treatment of many benign or malignant diseases of the vocal cords and allows bimanual surgery of the endolarynx (Larner et al., 2019). In suspension laryngoscopy, a significant force is exerted on the tongue and neck tissues due to the abutment mechanism used to visualize the larynx and pharynx, which are located deeper than the oral cavity. This force causes symptoms such as sore throat, dysphagia, paresis, cough, taste disorder, oral injury, and hoarseness in the postoperative period (Larner et al., 2019; Tsang et al., 2020; Taliercio et al., 2017).In the literature, it has been reported that patients experience sore throat, cough, dysphagia, and hoarseness symptoms after suspension laryngoscopy (Larner et al., 2019; Taliercio et al., 2017; Okui et al., 2020). Pharmacological and non-pharmacological methods can be applied to prevent sore throat and dysphagia after suspension laryngoscopy. The interventions that start while the patient is still in the recovery room to prevent postoperative sore throat and swallowing difficulties are the responsibility of the recovery unit nurses. Being aware of the problems such as sore throat and swallowing difficulties experienced by patients after suspension laryngoscopy, effective nursing practices should be developed to prevent these problems and their possible consequences. Therefore, the aim of this study is to examine the effect of cold vapor on sore throat and dysphagia in the early postoperative period after suspension laryngoscopy.

DETAILED DESCRIPTION:
Suspension laryngoscopy (SL) is a surgical procedure that is widely applied in the diagnosis and treatment of many benign or malignant diseases of the vocal cords and allows bimanual surgery of the endolarynx (Larner et al., 2019).In order to prevent any pain and gag reflex, the patients are placed in the supine position, neck hyperextension and head supported position on the operating table for the intervention performed under general anesthesia. With this position, it is aimed to place the microlaryngoscope and to ensure the patient's throat opening (Tsang et al., 2020; Taliercio et al., 2017).

In suspension laryngoscopy, a significant force is exerted on the tongue and neck tissues due to the abutment mechanism used to visualize the larynx and pharynx, which are located deeper than the oral cavity. This force causes symptoms such as sore throat, dysphagia, paresis, cough, taste disorder, oral injury, and hoarseness in the postoperative period (Larner et al., 2019; Tsang et al., 2020; Taliercio et al., 2017).In a study examining the complications experienced by patients after suspension laryngoscopy in the literature, Okui et al. reported that 66% of the patients experienced at least one complication, the most common complication was sore throat with 40%, and tongue numbness with 13.8%, cough with 13.4%, oral injuries with 11.5%, and taste disorders with 11.5% (Okui et al., 2020). In another study, it was reported that the most common postoperative complaints after suspension laryngoscopy were sore throat in 29% and hoarseness in 23% of the patients, while other less common symptoms were cough, frequent throat clearing, intermittent ear pain, and globus sensation (Larner et al., 2019). In another study, it was reported that 76% of the patients described a sore throat that continued for 3 days after the surgery, and that 36% of them continued after the 3rd day after the surgery (Taliercio et al., 2017).

Pharmacological analgesic agents are frequently used to relieve symptoms of sore throat and dysphagia that occur in patients after suspension laryngoscopy (Jung and Kimm, 2013; Paltura et al., 2020). In the literature, there are many studies on the successful application of non-pharmacological agents in the treatment of pain (Bulut et al., 2016; Şahbaz and Khorshid, 2020; Zaman and Karahan, 2020; Guidelenes on the Management of Postoperative Pain, Management of Postoperative Pain, 2016). Patients with post-operative throat complaints are recommended practices that reduce complaints such as taking warm liquids, not taking solid food, sucking ice chips, using lozenges, and applying steam.

The cold application creates vasoconstriction in the vessels in the area where it is applied, decreases the metabolic rate, and reduces edema. The cold application reduces muscle temperature by reducing the tension sensitivity of muscle spindles with the reflex effect of heat receptors or inactivating trigger points in the muscles and helps to reduce muscle spasm. Thus, it decreases skin sensitivity by lowering the temperature of nerve fibers and receptors. Cold application is especially useful in post-traumatic pain, swelling, and muscle spasm. Although it is seen that pharmacological, non-pharmacological, and herbal methods are applied to reduce postoperative sore throat and dysphagia in the literature, no study has been found examining the effect of cold vapor on sore throat and dysphagia. Therefore, the aim of this study is to examine the effect of cold vapor on sore throat and dysphagia in the early postoperative period after suspension laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* To undergo suspension laryngoscopy
* Having an ASA score of 1-2 points
* Not having any respiratory problems before the operation
* Not having a neurological disease related to swallowing
* Not having a sore throat due to cancer and chronic diseases
* Having a Modified Mallampati score of 1-2 points
* Getting 2 points from the Ramsay Sedation scale in the postoperative recovery room
* Having a Modified Aldrete score of at least 9 points in the postoperative recovery room
* The duration of the operation is at least 30 minutes
* To be willing to participate in the study.

Exclusion Criteria:

* To undergo emergency surgery
* Being under the age of 18
* Having an ASA score of 3 and above
* Having any respiratory problems in the preoperative period
* Having a neurological disease related to swallowing
* Having a sore throat due to cancer and chronic diseases
* Having a Modified Mallampati score of 3 or higher
* The duration of the operation is less than 30 minutes
* Not agreeing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-21 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Cold vapor | First 24 hours after surgery
  The Visual Analogue Scale (VAS) of the patients for sore throat who underwent cold vapor is decreased compared to those who do not. A score between 0 and 10 is taken from the VAS. It is good that the score from the VAS has decreased.
Cold vapor | First 24 hours after surgery
  The Numeric Rating Scale (RTS) of the patients for dysphagia who underwent cold vapor is decreased compared to those who do not. A score between 0 and 10 is taken from the RTS. It is good that the score from the RTS has decreased.

IPD SHARING:
Plan to Share IPD: Undecided
A decision will be made after consultation with other researchers.

REFERENCES:
- [Background] Larner SP, Fornelli RA, Griffith SD. Consistent Technique Limits Suspension Laryngoscopy Complications. Int Arch Otorhinolaryngol. 2019 Jul;23(3):e305-e310. doi: 10.1055/s-0039-1684036. Epub 2019 May 28. PMID 31360250
- [Background] Tsang TM, Brett O, Hu A. Patient Perception and Duration of Pain after Microdirect Laryngoscopy. Otolaryngol Head Neck Surg. 2020 May;162(5):702-708. doi: 10.1177/0194599820907904. Epub 2020 Mar 10. PMID 32151190
- [Background] Taliercio S, Sanders B, Achlatis S, Fang Y, Branski R, Amin M. Factors Associated With the Use of Postoperative Analgesics in Patients Undergoing Direct Microlaryngoscopy. Ann Otol Rhinol Laryngol. 2017 May;126(5):375-381. doi: 10.1177/0003489417693862. Epub 2017 Feb 1. PMID 28397564
- [Background] Okui A, Konomi U, Watanabe Y. Complaints and Complications of Microlaryngoscopic Surgery. J Voice. 2020 Nov;34(6):949-955. doi: 10.1016/j.jvoice.2019.05.006. Epub 2019 May 31. PMID 31160183
- [Background] Jung H, Kim HJ. Dexamethasone contributes to the patient management after ambulatory laryngeal microsurgery by reducing sore throat. Eur Arch Otorhinolaryngol. 2013 Nov;270(12):3115-9. doi: 10.1007/s00405-013-2708-5. Epub 2013 Sep 22. PMID 24057101
- [Background] Paltura C, Guvenc A, Develioglu ON, Yelken K, Kulekci M. Original Research: Aerosolized Lidocaine: Effective for Safer Arousal After Suspension Laryngoscopy. J Voice. 2020 Jan;34(1):130-133. doi: 10.1016/j.jvoice.2018.08.012. Epub 2018 Sep 15. PMID 30227980
- [Background] Bulut H, Erden S, Demir SG, Cakar B, Erdogan Z, Demir N, Ay A, Aydin E. The Effect of Cold Vapor Applied for Sore Throat in the Early Postoperative Period. J Perianesth Nurs. 2016 Aug;31(4):291-7. doi: 10.1016/j.jopan.2014.10.005. Epub 2016 Feb 24. PMID 27444760
- [Background] Sahbaz M, Khorshid L. The Effect of Cold Vapor and Ice Cube Absorption in the Early Postoperative Period on Sore Throat and Hoarseness Induced by Intubation. J Perianesth Nurs. 2020 Oct;35(5):518-524. doi: 10.1016/j.jopan.2019.12.007. Epub 2020 May 10. PMID 32402773
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- See also: Zaman, F. & Karahan, E. (2020). Effect of Cold Vapor Treated to Thyroidectomy Patients During Early Postoperative Period, East J Med 25(1): 118-125, DOI: 10.5505/ejm.2020.18189 — https://jag.journalagent.com/ejm/pdfs/EJM-18189-ORIGINAL_ARTICLE-KARAHAN.pdf